CLINICAL TRIAL: NCT00118794
Title: Randomized Trial of the Safety and Effectiveness of Lapdap and Coartemether for Uncomplicated Malaria in Operational Settings
Brief Title: Lapdap and Coartemether for Uncomplicated Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council (Other Government); National Malaria Control Programme, The Gambia (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCC975; SCC975
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2006-02-01 (Estimated); Status verified 2005-01

CONDITIONS: Malaria
Keywords: uncomplicated malaria; G6PD deficiency; haemolytic anaemia; Lapdap; Artemsinin based combination treatment; compliance; pragmatic trials
MeSH Terms: conditions — Malaria; Glucosephosphate Dehydrogenase Deficiency; Anemia, Hemolytic; Patient Compliance | interventions — chloroguanil, dapsone drug combination; Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: Chlorproguanil-dapsone (Lapdap)
Drug: Lumefantrine-artemether (Coartemether )

SUMMARY:
Lapdap (chlorproguanil-dapsone) is an affordable and effective drug, but patients with glucose-6-phosphate dehydrogenase (G6PD) A- deficiency are more susceptible to the haemolytic effects of the dapsone component of Lapdap; therefore there is a need to evaluate the extent to which the risks associated with the use of the drug in settings without G6PD screening might outweigh the benefits to malaria treatment. The investigators will evaluate, in operational settings, the safety and effectiveness of Lapdap and coartemether (lumefantrine-artemether) for treatment of uncomplicated malaria in patients 6 months to 10 years of age.

DETAILED DESCRIPTION:
Patients with uncomplicated malaria will be recruited at three health centres in the Gambia. Children aged 6 months to 10 years presenting with a history of illness, who have a fever or recent history of fever, will be screened; those with uncomplicated malaria, a positive blood smear with a parasite density of 500 to 200,000 parasites/µl, monoinfection with P. falciparum, and a packed cell volume of >=20%, will be invited to enroll into the study and if consent is given, will be randomized to receive three daily doses of lapdap, or a six-dose course of Coartem. The first dose will be given by the mother under direct observation by the dispensing nurse; subsequent doses will be given at home unsupervised. Children will be followed up actively three times; on day 3, to assess adherence to the treatment regimen, and on days 14 and 28, to assess parasitological and haematological recovery. The mother/caregiver of the child will be encouraged to bring the child to the clinic if the child does not improve or if she is concerned about the child's health. On day 3, the parent/caregiver will be visited at home (after the last dose should have been taken) in order to check for any leftover medication, and to ask about compliance and adverse reactions. A finger prick blood sample will be taken for Hb measurement by haemocue in the field and for a filter paper sample for measurement of drug concentration. The investigators will employ a longitudinal randomized design, whereby subsequent episodes of malaria will be treated according to the original randomization. This will enable better assessment of cumulative effects of repeated treatments on anaemia and on tolerability. Since patients with glucose-6-phosphate dehydrogenase (G6PD) A- deficiency are more susceptible to the haemolytic effects of the dapsone component of Lapdap, the investigators will determine the G6PD genotype and enzymatic activity, in order to evaluate the extent to which the risks associated with the use of the drug in settings without G6PD screening might outweigh the benefits to malaria treatment.

ELIGIBILITY:
Inclusion Criteria:

* presentation at health centre with febrile illness
* monoinfection with P falciparum
* parasitaemia >=500/microlitre
* fever or history of fever

Exclusion Criteria:

* signs of severe or complicated malaria (persistent vomiting with or without dehydration, history of convulsion during the present illness, inability to sit or stand, parasitaemia >200,000/ul)
* severe malnutrition
* clinically evident concomitant disease
* PCV <20%
* history of allergy to the study medications
* residence outside the study area and hence difficult to follow up

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200
Dates: Start 2004-09; Study Completion 2005-06

PRIMARY OUTCOMES:
Clinical failure by day 28

SECONDARY OUTCOMES:
Incidence of severe anaemia by day 28
Compliance
Incidence of adverse events
Parasitological failure by day 28
Clinical and parasitological failure rates by day 14
Fall in Hb of 2g/dl or more from screening value

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Milligan, BSc MSc PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Sam K Dunyo, MD PhD, Principal Investigator — Medical Research Council
Locations (1):
- Medical Research Council Laboratories, Banjul, City of Banjul, The Gambia

REFERENCES:
- [Derived] Dunyo S, Sirugo G, Sesay S, Bisseye C, Njie F, Adiamoh M, Nwakanma D, Diatta M, Janha R, Sisay Joof F, Temple B, Snell P, Conway D, Walton R, Cheung YB, Milligan P. Randomized trial of safety and effectiveness of chlorproguanil-dapsone and lumefantrine-artemether for uncomplicated malaria in children in the Gambia. PLoS One. 2011;6(6):e17371. doi: 10.1371/journal.pone.0017371. Epub 2011 Jun 7. PMID 21666744